CLINICAL TRIAL: NCT05542758
Title: High-Intensity Interval Training: Impacts on Function, Neuromuscular Control, and Muscle Architecture
Brief Title: High-Intensity Interval Training for Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2003313
Record Dates: First submitted 2022-09-06; First posted 2022-09-15 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Age-Related Sarcopenia
Keywords: geriatrics; high-intensity interval training; rehabilitation

STUDY DESIGN:
Intervention Model Description: All participants will receive the 12-week high-intensity intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total Body HIIT Program (Experimental): This Total Body HIIT program (circuit and bike training) will involve 3 sessions per week (35-40 min on nonconsecutive days) progressed across the 12 weeks. All session will be lead by undergraduate exercise science students or doctor of physical therapy students and supervised by a physical therapist.
  Interventions: Other: Total Body HIIT Program

INTERVENTIONS:
Other: Total Body HIIT Program — One repetition maximums (1RM) and body weight (BW) will be recorded at prior to and at 6 weeks to tailor the program. The circuit will be completed twice during each session and the exercises will include: squats, medicine ball forward chest throws, medicine ball overhead throw, farmers walk, seated shoulder press, seated row sitting on a fitness ball, aerobic riser step-ups, foot ladder drills, and twisting medicine ball passes. The anaerobic component will be completed once during a session and on a stationary bike. The progression of exercise:rest seconds will be 20:40 for Weeks 1-4, 30:30 for Weeks 5-8, and 40:20 for Weeks 9-12. Each session will start with a 5 minute warm up and end with a 5-minute cool down. Participants will be given real time feedback about heart rate (goal range: 85-95% HRmax) and exercise movement velocity. Participants will be encouraged to surpass the velocity of the previous repetition.

SUMMARY:
This study will examine differences in a 12 week high-intensity interval training regimen. The Total Body HIIT program incorporates a resistance (circuit) and an anaerobic (bike) component in older adults. The specific objectives focus on examining cardiovascular endurance, neuromuscular function, and muscle architecture.

ELIGIBILITY:
Inclusion Criteria:

* 65-95 years of age or older
* Physical independent (Barthel Index)
* Physician clearance to participate
* No medication changes in previous 30 days
* No structured resistance training program in previous 6 months

Exclusion Criteria:

* Contraindications to high-intensity exercise39 (PAR-Q Questionnaire)
* Severe mental impairment (<18 on Montreal Cognitive Assessment)
* Neurodegenerative or acute neurological diagnoses (e.g., Parkinson's disease, stroke, traumatic brain injury)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in 6-Min Walk Test performance from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  The 6MWT will be assessed by tallying the number of laps a participant is able walk on a 100 ft straight path. Partially completed laps will be measured and added to the total distance. Participants will be allowed to take standing rest breaks, if necessary, but the time will continue during all rest breaks. Participants will be instructed to "cover as much ground as you can in 6 minutes".
Change in Voluntary Muscle Strength Tests (Isokinetics) from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Isokinetic strength testing on the hamstrings, quadriceps femoris, biceps brachii, and triceps brachii muscles at slow (60° per second), medium (180° per second), fast (300° per second) and fast unweighted (500° per second) speeds with three maximal repetitions performed for each speed to determine voluntary peak torque production capabilities at each speed using a dynamometer. During the strength testing assessments, each subject will be asked to push or pull "as hard as possible" against a lever arm on the dynamometer until the limb reaches the end of the range of motion.
Change in Voluntary Muscle Strength Tests (Isometrics) from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Isometric strength of the hamstrings, quadriceps femoris, biceps brachii, and triceps brachii muscles will be assessed using a dynamometer. For maximal voluntary isometric contraction assessments, participants will complete two, 3- to 4-second MVICs of the hamstrings, quadriceps femoris, biceps brachii, and triceps brachii. Participants will be instructed to "push or pull as hard and fast as possible" and hold against the dynamometer to achieve max voluntary torque and rate of torque development.
Change in Evoked Muscle Function Assessments: Evoked Peak Force from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Evoked muscle function will be assessed using electrical stimulation delivered to the superficial quadriceps femoris via a cathode-anode arrangement, with the cathode probe pressed into the femoral triangle over the femoral nerve and the anode fixed over the greater trochanter. Manual stepwise increases in stimulation will be completed until max contraction is achieved. Once max contraction is achieved, a maximal, single and doublet stimulus will be administered. The single stimulation will be used to elicit a max M-wave amplitude (defined as the max M-wave peak-to-peak amplitude). A doublet stimulus will be used to drive the muscle to maximal contraction capability to investigate the muscle contractile capability. To examine maximal contractile capacity, torque produced from the quadriceps femoris from the dynamometer during the first 50 ms, evoked peak force.
Change in Evoked Muscle Function Assessments: Evoked Peak Rate of Force Development from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Evoked muscle function will be assessed using electrical stimulation delivered to the superficial quadriceps femoris via a cathode-anode arrangement, with the cathode probe pressed into the femoral triangle over the femoral nerve and the anode fixed over the greater trochanter. Manual stepwise increases in stimulation will be completed until max contraction is achieved. Once max contraction is achieved, a maximal, single and doublet stimulus will be administered. The single stimulation will be used to elicit a max M-wave amplitude (defined as the max M-wave peak-to-peak amplitude). A doublet stimulus will be used to drive the muscle to maximal contraction capability to investigate the muscle contractile capability. To examine maximal contractile capacity, evoked peak rate of force development 0-50ms will be recorded resulting from a maximal doublet stimulus from the quadriceps femoris.
Change in Rate of Muscle Activation from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  To examine muscle activation, surface electromyographic (sEMG) signals collected during the voluntary and evoked muscle contractions will be collected from the quadriceps femoris (vastus lateralis, rectus femoris, and vastus medialis muscles), hamstrings (biceps femoris muscle), biceps brachii, and triceps brachii muscles. Peak muscle activation will be assessed as the peak sEMG amplitude. Rate of muscle activation will be assessed in the first 50 ms following muscle activation onset.
Change in Voluntary Electromechanical Delay from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  To examine muscle activation, surface electromyographic (sEMG) signals collected during the voluntary and evoked muscle contractions will be collected from the quadriceps femoris (vastus lateralis, rectus femoris, and vastus medialis muscles), hamstrings (biceps femoris muscle), biceps brachii, and triceps brachii muscles. Peak muscle activation will be assessed as the peak sEMG amplitude. Voluntary electromechanical delay will be calculated from the time difference from the onset of sEMG to the onset of force.
Change in Ultrasound-based Muscle Architecture: Cross-sectional Area from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Ultrasound images of the vastus lateralis, rectus femoris, biceps femoris, vastus medialis, biceps brachii, and triceps brachii will be obtained. Muscle cross-sectional area for each muscle will be assessed.
Change in Ultrasound-based Muscle Architecture: Echo Intensity from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Ultrasound images of the vastus lateralis, rectus femoris, biceps femoris, vastus medialis, biceps brachii, and triceps brachii will be obtained. Echo intensity for each muscle will be assessed.
Change in Muscle Biopsy-based Muscle Architecture from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Muscle biopsies will be collected to determine myofiber size from the quadriceps femoris (i.e., vastus lateralis). After necessary biopsy preparations, the distribution of myofiber type and size will be determined within each sample.

SECONDARY OUTCOMES:
Change in V02 peak from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Participants will complete a graded exercise test (2-min stages) on the cycle ergometer to evaluate VO2 peak. VO2 peak for each subject will be taken as the highest single VO2 value when at least two of the three following test criteria are satisfied: 1) A leveling off in VO2 despite an increase in power output, 2) maximal heart rate within 15 beats of age-predicted maximal heart rate (220-age), and 3) respiratory exchange ratio (RER) ≥1.1.
Change in Gait Speed from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Gait speed will be assessed with the 10-meter walk test (maximum comfortable walking speed).
Change in Functional Lower Body Strength from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Functional lower body strength will be assessed with the 5 times sit to stand test. This test requires participants to stand up and sit down 5 times without the use of upper extremities as fast as possible.
Change in Functional Upper Body Strength from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Functional upper body strength will be assessed with hand grip strength. Three repetitions of 30 second maximum hold on each hand will be completed.
Change in Balance: Center of Pressure Excursion from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Participants will statically stand on a force plate in three different scenarios (feet together eyes open, feet together eyes shut, and single-leg stance). Center of pressure excursion will be calculated to determine static balance.
Change in Balance: Functional Gait Assessment from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Participants will complete the functional gait assessment, a clinical assessment of walking ability under various conditions (e.g., stepping over an obstacle, walking backwards, etc.). Scores range from 0-30 with higher scores indicating better balance performance.
Change in Balance: Berg Balance Scale from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Participants will complete the Berg Balance Scale, a clinical assessment of static and dynamic balance abilities. The Berg Balance Scale Score ranges from 0-56 with higher scores indicating better balance performance.
Change in Health-Related Quality of Life from baseline to following HIIT intervention | change from baseline to immediately after the HIIT intervention
  Participants will complete the Short-Form Health Survey (SF-36) to assess health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be determined on a request case-by-case basis.